CLINICAL TRIAL: NCT02367755
Title: Combining Propofol With Therapeutic Hypothermia for Improving Survival and Neurological Prognoses in Patients Resuscitated From Cardiac Arrest
Brief Title: Therapeutic Hypothermia With Propofol in Survival and Neurological Prognoses After Cardiac Arrest
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yen-Wen Wu, Chief of Cardiology Division of Cardiovascular Medical Center and Department of Nuclear Medicine, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102060-F_102-FTN12
Record Dates: First submitted 2015-02-02; First posted 2015-02-20 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Hypothermia; Cardiac Arrest
Keywords: cardiopulmonary resuscitation; cardiac arrest; therapeutic hypothermia; propofol; lorazepam; cerebral perfusion; electroencephalography
MeSH Terms: conditions — Hypothermia; Heart Arrest | interventions — Propofol; Lorazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Experimental): propofol infusion at a rate of 3 mg/kg/hr during TH.
  Interventions: Drug: Propofol
- Lorazepam (Active Comparator): lorazepam infusion at a rate of 0.5 mg/kg/hr during TH.
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: Propofol — Propofol use during therapeutic hypothermia
  Other Names: P
  Arms: Propofol
Drug: Lorazepam — Lorazepam use during therapeutic hypothermia
  Other Names: L
  Arms: Lorazepam

SUMMARY:
Therapeutic hypothermia has been proven to significantly improve the survival and neurological prognoses in patients resuscitated from cardiac arrest. Propofol has been reported to exhibit potentials in mitigating ischemia-reperfusion injury via the antioxidative, anti-inflammatory and neuroprotective mechanisms. This study is to investigate the potentials of propofol in further improving the survival and neurological prognoses in this era of therapeutic hypothermia.

DETAILED DESCRIPTION:
Cardiac arrest and cardiopulmonary resuscitation (CPR) is a specific model of global ischemia/reperfusion (I/R) injury. Among all organ systems, brain is least tolerable to ischemic insult and I/R injury, which accounts for the usually poor survival and neurological outcomes in these patients even with initial success in resuscitation. Therapeutic hypothermia (TH) has been proven to significantly improve the survival and neurological prognoses in patients resuscitated from cardiac arrest. It has been recommended as a standard therapy in the post-resuscitation care since 2002. In the past few years, NTUH and FEMH have been actively promoted the application of TH in the post-resuscitation care, and both have achieved important progress. Based on these, the investigators seek to further improve the survival and neurological outcomes in this group of patients. Among the therapies with potential additive or synergistic protective mechanisms, propofol has been extensively studied, and shown to exhibit great potentials in mitigating ischemia-reperfusion injury via the antioxidative, anti-inflammatory and neuroprotective mechanisms. As sedatives are basic requirement during TH according to technical and ethical concerns, the combination of propofol and TH is not only justified but highly anticipated. The investigators therefore seek to investigate the potentials of propofol in further improving the survival and neurological prognoses in this era of therapeutic hypothermia.

Methods: This .is a prospective, single-blinded randomized clinical trial. The inclusion criteria include: (1) non-traumatic cardiac arrest (2) no regain of consciousness after return of spontaneous circulation (ROSC) (3) age >=20 years old and <= 90 years old. The exclusion criteria include (1) age < 20 y/o or > 90 y/o (2) pregnancy (3) traumatic cardiac arrest (4) fail to achieve ROSC (5) conscious recovery after ROSC (6) contraindications for TH, such as massive bleeding, infections, etc (7) terminal diseases (8) conscious disturbance before cardiac arrest (9) fail to obtain informed consent (10) families refuse to undergo clinical trial. The study will be divided to two groups: (1) Lorazepam group: lorazepam infusion at a rate of 0.5 mg/kg/hr during TH. (2) Propofol group: propofol infusion at a rate of 3 mg/kg/hr during TH. The primary endpoints will be (1) survival (2) neurological outcomes as indicated by cerebral performance category (CPC) scale. The secondary endpoints include (1) 99mTc ECD scan (perfusion and viability), (2) clinical and EEG evidences of seizure. The blood pressure and heart rate will continuously monitored during TH and propofol/lorazepam infusion.

Expected Results: (1) Test if propofol further improves the survival and neurological outcomes in post-CPR patients undergoing TH (2) Test if propofol further improves cerebral perfusion and neuron viability in post-CPR patients undergoing TH (3) Test if propofol reduces the incidence and severity of seizures post-CPR, (4) Test if propofol significantly influence hemodynamics when combined with TH Clinical Implications: Propofol is a clinically available sedative agent. If this trial demonstrates that propofol further improves the survival and neurological outcomes in post-resuscitation patients undergoing TH, it would become an important evidence justifying implementation in clinical practice

ELIGIBILITY:
Inclusion criteria:

1. non-traumatic cardiac arrest
2. no regain of consciousness after return of spontaneous circulation (ROSC)
3. age >=20 years old and <= 90 years old.

Exclusion criteria:

1. age < 20 y/o or > 90 y/o
2. pregnancy
3. traumatic cardiac arrest
4. fail to achieve ROSC
5. conscious recovery after ROSC
6. contraindications for TH, such as massive bleeding, infections, etc
7. terminal diseases
8. conscious disturbance before cardiac arrest
9. fail to obtain informed consent
10. families refuse to undergo clinical trial
11. allergy to propofol or lorazepam.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Neurologic statue at discharge | at dicharge
  Glasgow score, cerebral performance category scale

SECONDARY OUTCOMES:
Brain SPECT The standard 99mTc-ethylene L-cysteinate dimer [ECD] will be done on day 5-14 post-resuscitation. The perfusion will be assessed, and the viability of the cerebral tissue will be interpreted using SPECT, by 2 experienced nuclear m | day 5-14 post-resuscitation
  Regional Scores of Tc-99m ECD Brain SPECT
From ROSC to recovery of consciousness | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Recovery of consciousness: being able to follow orders. participants will be followed for the duration of hospital stay, an expected average of 4 weeks.
Survival to discharge | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Wen Wu, MD, PhD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Not share data